CLINICAL TRIAL: NCT07069946
Title: Effect of Weight Bearing Exercises With Neuromuscular Electrical Stimulation on Balance and Functional Abilities In Children With Hemiplegia
Brief Title: Weight Bearing Exercises With NMES on Balance and Functional Abilities In Children With Hemiplegia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdulrahman Ahmad Mohamad Mostafa, Abdulrahman Ahmad Mohamad Mostafa, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No:P.T.REC/012/005783
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: weight-bearing exercises program; neuromuscular electrical stimulation; balance; functional abilities; hemiplegic cerebral palsy

STUDY DESIGN:
Intervention Model Description: weight-bearing exercise and neuromuscular electrical stimulation
Who Masked: Outcomes Assessor
Masking Description: sealed envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): This group will include 15 children with hemiplegic cerebral palsy and will receive a split 60 minutes, 30 minutes of traditional physical therapy and 30 minutes of weight-bearing exercise , 3 sessions/ week for 8 weeks.
  Interventions: Other: traditional physical therapy and weight-bearing exercise
- Study group (Experimental): This group will include 15 children with hemiplegic cerebral palsy and will receive the same 60 minutes session of the control group in addition to neuromuscular electrical stimulation during the 30 minutes weight-bearing program , 3 sessions/ week for 8 weeks.
  Interventions: Other: neuromuscular electrical stimulation , traditional physical therapy and weight-bearing exercise

INTERVENTIONS:
Other: traditional physical therapy and weight-bearing exercise — They will receive 60 minute session, 3 times/ week for 8 weeks as following:
  * 30 minutes of traditional physical therapy program : Includes: Strengthening, Stretching, Balance, Postural Control, Functional Mobility and Gait Training.
  * 30 minutes of seven different weight-bearing exercises program of exercises with three of those being repeated on the left and right sides to make a total of ten exercises, each held for 3 minutes, the exercises include: hamstring stretch, calf stretch, half kneeling balance, static squat, bridge, four point kneeling and four point kneeling with leg extension the exercises include: : Hamstring stretch,Calf stretch , Half kneeling balance , Static Squat, Bridge, Four point kneeling with leg extension, and Four point kneeling.
  Arms: Control group
Other: neuromuscular electrical stimulation , traditional physical therapy and weight-bearing exercise — They will receive 60 minute session, 3 times/ week for 8 weeks as following:
  * 30 minutes of the same traditional physical therapy as the control group.
  * 30 minutes of the same weight-bearing exercises program as the control group adding to it the neuromuscular electrical stimulation on: Tibialis anterior, Quadriceps, Paraspinal muscles.
  * NMES Parameters :
    * Device: Everyway-EV-906.
    * Frequency: 30-35 Hz (to optimize muscle endurance and motor unit recruitment).
    * Pulse Width: 250-300 µs.
    * Intensity: Adjusted to elicit visible muscle contraction without discomfort (submaximal, (25-30 mA).
    * Electrode Placement:
      * Lower Limb: Tibialis anterior (for dorsiflexion) and quadriceps (for knee stability) during weight-bearing (El-Shamy and El Kafy, 2021).
      * Trunk: Paraspinal muscles (for postural control) during static squats and bridging
  Arms: Study group

SUMMARY:
This study will be conducted to investigate the combining effect of weight-bearing exercises program with neuromuscular electrical stimulation on balance and functional abilities in children with hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
Hemiplegic cerebral palsy (HCP) is characterized by unilateral motor impairment, with the upper extremities typically exhibiting greater functional limitations compared to the lower limbs. This subtype constitutes approximately 20-30% of cerebral palsy cases and arises from unilateral injury to the developing brain, resulting in asymmetrical muscle tone abnormalities, joint deformities, and restricted range of motion. Individuals with HCP often display irregular, uncoordinated movements on the affected side, significantly impacting motor performance. Children with spastic hemiplegia experience decreased balance ability and abnormal gait because of decreased weight-bearing in the paretic leg. Diminished motor ability in the paretic leg causes weakening of the quadriceps, ankle plantar flexors, and ankle dorsiflexors.

The rehabilitation of balance and walking ability is crucial for children diagnosed with cerebral palsy. Weight-bearing exercises are defined as physical activities in which the feet and legs support the body's weight while moving against gravity. These exercises are essential for stimulating bone growth, improving bone density, and enhancing musculoskeletal health. Examples of weight-bearing exercises include walking, running, jumping, dancing, climbing stairs, playing sports such as soccer or basketball, and engaging in recreational activities like hiking or skating. Regular participation in weight-bearing exercises is particularly important for children and adolescents, as it helps maximize peak bone mass during growth and reduces the risk of osteoporosis later in life.

Exercise programs for cerebral palsy exhibit significant variation in terms of their types, such as gait training, body-weight-supported treadmill training, balance training, or multi-component approaches, and the efficacy of different exercises has not been established in improving the functional abilities of children with cerebral palsy. Studies suggest that integrating neuromuscular electrical stimulation (NMES) with conventional rehabilitation approaches enhances therapeutic outcomes compared to using NMES in isolation .

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with hemiplegic cerebral palsy.
* Their age will range from 6-10 years.
* Both sexes will be included.
* All participants will be able to follow simple commands.
* They will be graded as mild spasticity of the lower limbs according to MAS grade 1 to 1+ .
* They will be at levels I and II based on the GMFCS

Exclusion Criteria:

* Children with any neurological conditions other than hemiplegic cerebral palsy will be excluded from the study.
* Musculoskeletal problems or congenital deformity.
* Children with fixed contracture.
* Lower limb surgery in the last one year.
* Rhizotomy, or injection of botulinum toxin into the lower limb muscles during the previous 6 months.
* Receive any medications that affect the arousal and alertness status.
* Children having epilepsy.
* Visual or auditory defects.
* Skin sensitivity.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Balance | up to 8 Weeks
  The HUMAC Balance System (HUMAC2015® Version: 15.000.0103; Computer Sports Medicine, Inc.) will assess pediatric postural balance before and after treatment. This system, featuring a force plate and specialized software, provides precise and reliable measurements of static and dynamic balance, supported by established reliability in pediatric studies.

SECONDARY OUTCOMES:
The Gross Motor Function Measure GMFM | Up to 8 weeks
  The GMFM Will be used for functional abilities evaluation for all children participating in the study before and after treatment procedures. Including the 88-item (GMFM-88) and 66-item (GMFM-66) versions, assesses gross motor function changes in children with cerebral palsy. Both demonstrate high validity and reliability . An adapted GMFM-88 version shows excellent test-retest and inter observer reliability

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman Mostafa, MSc., Principal Investigator — Master degree